CLINICAL TRIAL: NCT04856228
Title: Ultrasonographic and Electrophysiological Evaluation of The Presence of Radial Tunnel Syndrome in Patients With Resistant Lateral Epicondylitis
Brief Title: Radial Tunnel Syndrome in Resistant Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aslinur Keles Ercisli, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-83045809-604.01.02-7933
Record Dates: First submitted 2021-04-16; First posted 2021-04-23 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Radial Tunnel Syndrome; Lateral Epicondylitis; Radial Nerve Compression; Epicondylitis of the Elbow
Keywords: radial nerve; radial tunnel syndrome; lateral epicondylitis; ultrasonography; electrophysiology
MeSH Terms: conditions — Radial Neuropathy; Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic single group (Other): Patients diagnosed with lateral epicondylitis with physical examinations will be evaluated with electrophysiology After electrophysiological evaluations, patients' effected extremity evaluated with ultrasonography for lateral epicondylitis and radial tunnel syndrome and compared with uneffected side 30 minutes after posterior interosseous nerve block with 1 cc 2% lidocaine with USG guide, full examination will be repeated for evaluation of NRS score changing to exact diagnose of radial tunnel syndrome 30 minutes after lateral epicondyle 1 cc 2% lidocaine injection with USG guide, full examination will be repeated for evaluation of NRS score changing to final diagnose of lateral epicondylitis
  Interventions: Diagnostic Test: diagnostic posterior interosseous nerve lidocaine injection

INTERVENTIONS:
Diagnostic Test: diagnostic posterior interosseous nerve lidocaine injection — ultrasound guided posterior interosseous nerve and lateral epicondyle 1 ml 2% lidocaine injection
  Other Names: diagnostic lateral epicondyle lidocaine injection

SUMMARY:
Lateral elbow pain can be difficult to diagnose because of the different pathologies or combinations of pathologies that can cause this clinic. Although lateral epicondylitis is the most common cause of lateral elbow pain, symptoms of radial tunnel syndrome may masquerade as lateral epicondylitis or they can be seen together with rate of 21-41%. The aim of the study is; to evaluate the presence of radial tunnel syndrome in the patients who have resistant lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE), also known as "tennis elbow," is an overuse syndrome of the common extensor tendon (CET), predominantly affecting the extensor carpi radialis brevis. History and physical examination including manual provocation tests are key elements for the diagnosis.

Ultrasound imaging of the CET is an important complementary method to the clinical diagnosis of LE. It provides information about the severity of the disease with evidence of tendon thickening, focal/diffuse areas of decreased echogenicity in the tendon, epicondylar cortical irregularity or spur formation, and increased vascularity in case of local inflammation depicted by power- Doppler imaging.

Radial tunnel syndrome (RTS) is a dynamic/intermittent compression neuropathy of the radial nerve, where different structures can potentially compress the nerve. Local inflammatory and/or vascular changes (scarring, fibrosis), which are seen in LE may lead to compression of the radial nerve or its branches (especially the deep branch) at the radial tunnel. While RTS can often be the cause of refractory LE, some patients with LE actually have RTS concomitantly. The diagnosis of RTS is difficult/controversial due to inconclusive findings on electrophysiological tests and its close relationship with LE. Ultrasound is a superior imaging modality that can be used as an adjunct to electromyography for the evaluation of peripheral nerve problems. It can be used to diagnose compression neuropathies and to identify the entrapment site of the nerve. For the exact diagnosis of RTS complete relief should be achieved with a nerve block at the radial tunnel. Patients who have RTS coexisting with LE (18-43%) usually experience incomplete relief.

The purpose of the study is; to evaluate the RTS and LE with physical examination, special clinical tests, electrophysiological and ultrasonographic examinations and, to confirm the presence of RTS accompanying LE with the evaluation of clinical findings after the posterior interosseous nerve and lateral epicondyle diagnostic injections.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Had persistent lateral elbow pain at least 6 months' duration with suspected lateral epicondylitis
3. Be able to understand enough Turkish to complete the outcome questionnaire
4. Patients whose informed consent was obtained for paticipation in the study

Exclusion Criteria:

1. Fibromyalgia
2. History of surgery in the elbow
3. History of fracture that cause the deformity at radius/ulna
4. Pregnancy or breastfeeding
5. Inflammatuar arthropathy in upper extremities
6. Osteoarthritis in the upper extremities
7. Neurological disabilities that effect the upper extremity functions
8. Cervical radiculopathy that effect the level of C6-C7

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain via Nurmerical Rating Scale at 30 Minutes after PIN/Lateral Epicondyle Injection | Baseline, 30 minutes after PIN injection, 30 minutes after lateral epicondyle injection
  Pain of the participants will be assessed by one of the most commonly used pain scale "numerical rating scale". It is numeric version of visual analog scale in which a patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine". Participant is asked to indicate rates of their pain on the day of presentation during resting, during function and physical examination as a baseline and, 30 minutes after PIN injection for each, 30 minutes after lateral apicondyle injection for each.

SECONDARY OUTCOMES:
Grip strength via dynamometer | Baseline
  Handgrip strength was measured by using a Jamar Hand Dynamometer with patients seated, their elbow by their side and flexed to right angles, and a neutral wrist position. Three measurements were performed for both side, and the mean score was recorded (effected site and dominancy were noted)
The Patient-Rated Tennis Elbow Evaluation (PRTEE) | Baseline
  PRTEE is a validated pain severity and functional disability scale that assesses pain (5 questions graded 0 to 10) and functional disability (10 questions graded 0 to 10). Functional scores are then halved and added to pain scores. The minimum score is 0 (no pain or disability) and the maximum is 100 (severe pain and disability)
Disabilities of Arm, Shoulder, and Hand (DASH) Questionnaire | Baseline
  The DASH is a validated questionnaire designed to measure upper limb disability and symptoms. Functional domains include physical, social, and psychological. It uses a single-scale, 30-item questionnaire of upper extremity function and symptoms. The minimum sum score is 30 points; the maximumscore is 150 points
The 36-Item Short Form Health Survey Questionnaire (SF-36) | Baseline
  SF-36 is a popular instrument for evaluating Health-Related Quality of Life and commonly used, general health assessment that is reliable and valid for overall outcome. It measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Ulku Akarirmak, Study Director — Istanbul University - Cerrahpasa; Aslinur Keles Ercisli, Principal Investigator — Istanbul University - Cerrahpasa; Deniz Palamar Kadioglu, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekstrom RA, Holden K. Examination of and intervention for a patient with chronic lateral elbow pain with signs of nerve entrapment. Phys Ther. 2002 Nov;82(11):1077-86. PMID 12405872
- [Background] Ritts GD, Wood MB, Linscheid RL. Radial tunnel syndrome. A ten-year surgical experience. Clin Orthop Relat Res. 1987 Jun;(219):201-5. PMID 3581572
- [Background] Newcomer KL, Martinez-Silvestrini JA, Schaefer MP, Gay RE, Arendt KW. Sensitivity of the Patient-rated Forearm Evaluation Questionnaire in lateral epicondylitis. J Hand Ther. 2005 Oct-Dec;18(4):400-6. doi: 10.1197/j.jht.2005.07.001. PMID 16271686
- [Background] Tran N, Chow K. Ultrasonography of the elbow. Semin Musculoskelet Radiol. 2007 Jun;11(2):105-16. doi: 10.1055/s-2007-1001876. PMID 18095243
- [Background] Gurcay E, Karaahmet OZ, Kara M, Onat SS, Ata AM, Unlu E, Ozcakar L. Ultrasonographic Evaluation of the Radial Nerves in Patients with Unilateral Refractory Lateral Epicondylitis. Pain Med. 2017 Mar 1;18(3):396-402. doi: 10.1093/pm/pnw181. PMID 27477582